CLINICAL TRIAL: NCT02308228
Title: Novel Actions of Metformin to Augment Resistance Training Adaptations in Older Adults
Brief Title: Metformin to Augment Strength Training Effective Response in Seniors (MASTERS)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Philip Kern (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor-Investigator, Philip Kern, M.D., University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1R01AG046920-01A1 (NIH)
Record Dates: First submitted 2014-11-25; First posted 2014-12-04 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-08

CONDITIONS: Aging
Keywords: Aging; Hypertrophy; Metformin; Strength; Muscle
MeSH Terms: conditions — Hypertrophy | interventions — Resistance Training; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Participants will be randomized to receive Metformin (1700 mg/day) for a period of 16 weeks; 2 weeks of Metformin only followed by 14 weeks of continued Metformin use in combination with progressive resistance training.
  Interventions: Behavioral: Progressive Resistance Training; Drug: Metformin
- Placebo, Sugar Pill (Placebo Comparator): Participants will be randomized to receive placebo sugar pills (1700 mg/day) for a period of 16 weeks; 2 weeks of placebo only followed by 14 weeks of continued placebo use in combination with progressive resistance training. Placebos will be almost identical to the Metformin medication.
  Interventions: Behavioral: Progressive Resistance Training

INTERVENTIONS:
Behavioral: Progressive Resistance Training — Participants will complete 14 weeks (42 sessions, 3x/week) of progressive resistance training which will consist of 8 constant load movements to train all major muscle groups bilaterally.
  Other Names: Strength Training
Drug: Metformin — Participants will be randomized to receive metformin in conjunction with their strength training program.
  Other Names: Glucophage XR
  Arms: Metformin

SUMMARY:
The purpose of this study is to determine whether a commonly prescribed drug, metformin, can enhance the benefits seen during resistance exercise such as increased muscle mass and strength.

DETAILED DESCRIPTION:
Muscle mass and strength are critical determinants not only of a person's quality of life and functional independence, but also metabolic health, as muscle is the organ primarily responsible for insulin-mediated glucose uptake. The elderly suffer obligatory losses of muscle mass and strength, exacerbated by illness and physical inactivity. Progressive resistance exercise training (PRT) is the most effective intervention identified to improve muscular strength, and combat the muscle atrophy of aging (sarcopenia); however, overall the muscle response to PRT is blunted in the elderly and variability of response increased, with some individuals actually losing muscle mass. The Bamman and Peterson labs have independently been studying the molecular and cellular mechanisms underlying the "non-responder" phenotype, with the goal of identifying novel intervention strategies to promote mass and strength gains to improve function. We hypothesize that the abundance of anti-inflammatory, alternatively activated M2 macrophages in muscle predicts response to PRT in the elderly; those with the highest number of M2 macrophages and lowest inflammatory gene expression prior to the start of training gained the most mass. Further, we determined that metformin treatment increased M2 macrophage abundance, and decreased inflammatory cytokine gene expression. These provocative findings have led us to our central hypothesis that adjuvant metformin may improve the responses to PRT in the elderly by altering the muscle tissue inflammatory environment, thereby enhancing mechanisms that drive PRT-induced myofiber hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age.
* Independently mobile with a SPPB score 3-12.
* Access to transportation.
* Capable of providing informed consent (cognitively intact).

Exclusion Criteria:

* Obesity (BMI>30)
* Serum creatinine >1.4 because of risk of lactic acidosis with metformin.
* History of regular resistance training within the past year.
* History (or ECG evidence) of previous myocardial infarction, history of congestive heart failure.
* Current angina pectoris or symptoms of myocardial ischemia or congestive heart failure.
* Chronic aspirin or NSAID use (unless it can be safely stopped prior to the biopsies), and any other use of an anticoagulant (e.g., Coumadin) or history of bleeding.
* History of alcoholism or liver disease.
* History of hypo- or hyper-coagulation disorders including subjects taking Coumadin.
* Any end-stage disease and/or a life expectancy less than one year.
* Neurological, musculoskeletal, or other disorder that would preclude them from completing resistance training and all performance tests.
* Uncontrolled hypertension.
* Diabetes mellitus as demonstrated with- HgbA1C>6.5, or fasting glu>126 mg/dl.
* Any other medical condition that would interfere with testing or increase one's risk of complications during exercise, as judged by the study physicians.
* Any other condition or events considered exclusionary by the PI and/or physician, such as non-compliance.
* Lidocaine allergy (1% lidocaine is the local anesthetic used during the muscle biopsy procedure).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Peterson, Ph.D., Principal Investigator — University of Kentucky; Philip Kern, M.D., Principal Investigator — University of Kentucky; Marcas Bamman, Ph.D, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long DE, Kosmac K, Dungan CM, Bamman MM, Peterson CA, Kern PA. Potential Benefits of Combined Statin and Metformin Therapy on Resistance Training Response in Older Individuals. Front Physiol. 2022 Apr 14;13:872745. doi: 10.3389/fphys.2022.872745. eCollection 2022. PMID 35492586
- [Derived] Long DE, Peck BD, Tuggle SC, Villasante Tezanos AG, Windham ST, Bamman MM, Kern PA, Peterson CA, Walton RG. Associations of muscle lipid content with physical function and resistance training outcomes in older adults: altered responses with metformin. Geroscience. 2021 Apr;43(2):629-644. doi: 10.1007/s11357-020-00315-9. Epub 2021 Jan 18. PMID 33462708
- [Derived] Walton RG, Dungan CM, Long DE, Tuggle SC, Kosmac K, Peck BD, Bush HM, Villasante Tezanos AG, McGwin G, Windham ST, Ovalle F, Bamman MM, Kern PA, Peterson CA. Metformin blunts muscle hypertrophy in response to progressive resistance exercise training in older adults: A randomized, double-blind, placebo-controlled, multicenter trial: The MASTERS trial. Aging Cell. 2019 Dec;18(6):e13039. doi: 10.1111/acel.13039. Epub 2019 Sep 26. PMID 31557380
- [Derived] Long DE, Villasante Tezanos AG, Wise JN, Kern PA, Bamman MM, Peterson CA, Dennis RA. A guide for using NIH Image J for single slice cross-sectional area and composition analysis of the thigh from computed tomography. PLoS One. 2019 Feb 7;14(2):e0211629. doi: 10.1371/journal.pone.0211629. eCollection 2019. PMID 30730923
- [Derived] Long DE, Peck BD, Martz JL, Tuggle SC, Bush HM, McGwin G, Kern PA, Bamman MM, Peterson CA. Metformin to Augment Strength Training Effective Response in Seniors (MASTERS): study protocol for a randomized controlled trial. Trials. 2017 Apr 26;18(1):192. doi: 10.1186/s13063-017-1932-5. PMID 28441958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Number of individuals consented and further screened for eligibility = 144 Number of participants randomized to drug/placebo = 109 Number of participants completing exercise intervention with drug/placebo use = 94
Pre-assignment Details: Participants may have been excluded prior to randomization to study drug for the following reasons:
  1. Screen fail (OGTT, ECG, Blood results)
  2. Withdrawals (changed mind, lost to follow up, spouse screen fail)
Period: Overall Study
Arm/Group | Metformin | Placebo, Sugar Pill
Started | 54 | 55
Completed | 46 | 48
Not Completed | 8 | 7
Not completed — Adverse Event | 3 | 4
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo, Sugar Pill | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 53 | 53 | 106
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — Population: Data analyzed for those who completed the interventions = 94
  years
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 69.4 [66.8 to 72.3] | 69.3 [66.8 to 74.0] | 69.4 [66.8 to 73.2]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data analyzed for those who completed the interventions = 94
  Participants
    number analyzed (Participants) | 46 | 48 | 94
    Female | 22 | 29 | 51
    Male | 24 | 19 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data analyzed for those who completed the interventions = 94
  Participants
    number analyzed (Participants) | 46 | 48 | 94
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 46 | 48 | 94
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data analyzed for those who completed the interventions = 94
  Participants
    number analyzed (Participants) | 46 | 48 | 94
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 45 | 47 | 92
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 55 | 109
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Data analyzed for those who completed the interventions = 94
  kg/m^2
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 26.9 (3.1) | 25.7 (3.1) | 26.3 (3.1)
Short Physical Performance Battery (SPPB) [Mean (Inter-Quartile Range); unit: Scores on a Scale] — A physical performance measure based on balance, gait speed, and sit to stand. Total scores are provided as the sum of three subscales; 0-12 total range, 4-12 was required to be included in the study.
  Balance = 0-4 subscale Gait Speed = 0-4 subscale Sit to stand time = 0-4 subscale Higher scores = better overall performance Population: Data analyzed for those who completed the interventions = 94
  Scores on a Scale
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 11 [10 to 12] | 11 [11 to 12] | 11 [10.5 to 12]
Physical Activity Survey for the Elderly (PASE) [Median (Inter-Quartile Range); unit: Scores on a Scale] — Self Reported Physical Activity Score Median and inter-quartile ranges of the total activity score are reported. Total activity score is a sum of various domains including activity reported at home, during sports, housework, caring for other people, and work. The scale range is 0-793; higher scores indicate higher self-reported activity. Population: Data analyzed for those who completed the interventions = 94
  Scores on a Scale
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 155.5 [115.8 to 207.4] | 165.7 [133.4 to 210.5] | 159.3 [124.2 to 209.5]
Short Form-36 Physical Component (SF-36) [Median (Inter-Quartile Range); unit: Scores on a Scale] — Physical Function Component Norm Based Score Median and inter-quartile ranges of the physical function norm based score are reported as there is not a reported maximum.
  Questions related to physical function are scored 0-100. Physical function score = the average score of physical function questions. A z-score is calculated from the physical function score. The physical function norm based score is calculated from the physical function z-score.
  Scores above 50 would represent above average physical function where scores below 50 represent below average function. Population: Data analyzed for those who completed the interventions = 94
  Scores on a Scale
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 54.7 [49.1 to 57.5] | 55.2 [49.5 to 57.6] | 55.0 [49.1 to 57.6]
Short Form-36 Mental Component (SF-36) [Median (Inter-Quartile Range); unit: Scores on a Scale] — Mental Component Norm Based Score Median and inter-quartile ranges of the mental health norm based score are reported as there is not a reported maximum.
  Questions related to mental health are scored 0-100. Mental Health score = the average score of mental health questions. A z-score is calculated from the mental health score. The mental component norm based score is calculated from the mental health z-score.
  Scores above 50 would represent above average mental health where scores below 50 represent below average mental health. Population: Data analyzed for those who completed the interventions = 94
  Scores on a Scale
    number analyzed (Participants) | 46 | 48 | 94
    (all) | 56.7 [52.3 to 59.3] | 56.5 [54.6 to 59.1] | 56.6 [53.4 to 59.2]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Type 2 Myofiber Cross Sectional Area
Description: The ability of metformin to improve the hypertrophic response to resistance training will be determined. Muscle biopsies of the vastus lateralis will be used to quantify myofiber cross-sectional area. The percent change in type 2 myofiber size between week 16 and week 0 was used.
Time Frame: 16 weeks
Population: The largest, highest quality pairs of baseline and week 16 mounts were used for quantification of immunohistochemistry (N=30/group)
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Metformin | Placebo, Sugar Pill
Number analyzed (Participants) | 30 | 30
Percent change | 18.5 (31.5) | 14.5 (29.7)

2. Secondary Outcome: Percent Change in Normal Density Muscle Size by Computed Tomography
Description: The ability of metformin to improve the hypertrophic response at the whole muscle level will be quantified by computed tomography. Percent change in normal density muscle area will be calculated as the difference between week 16 and week 0.
Time Frame: 16 weeks
Population: Missing data points include those who, based on femur area, CT positioning at post measure was incorrect = 16. In addition, 1 subject was excluded from analysis as CT data indicated 45% loss of thigh muscle area, which was not consistent with other data for this subject.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Metformin | Placebo, Sugar Pill
Number analyzed (Participants) | 37 | 40
Percent change | 4.2 (9.1) | 10.5 (7.0)

3. Other Pre Specified Outcome: Percent Change in Muscle Strength
Description: Determine if metformin treatment augments strength gains in conjunction with progressive resistance training by one repetition maximum assessments. Maximum (1RM) leg extension muscle strength was assessed at week 4 (to account for neurological adaptations during the initial stages of the resistance program) and week 16. The percent change from week 4 to week 16 is reported.
Time Frame: Week 4 and week 16
Population: Some participants were not able to complete the procedure on the day of testing, injured etc
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Metformin | Placebo, Sugar Pill
Number analyzed (Participants) | 44 | 45
Percent change | 15.3 (18.5) | 23.1 (18.9)

4. Other Pre Specified Outcome: Percent Change in Total Body Lean Mass by DXA
Description: To determine if metformin improves changes in body composition associated with progressive resistance training. Percent change in total body lean mass in kg was calculated as the difference between week 16 and week 0 from a total body DXA scan.
Time Frame: 16 weeks
Population: Analysis of lean muscle mass for those who completed the interventions.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Metformin | Placebo, Sugar Pill
Number analyzed (Participants) | 46 | 48
Percent change | 0.41 (2.25) | 1.95 (2.69)

5. Other Pre Specified Outcome: Insulin Sensitivity
Description: A standard OGTT will be used to determine insulin sensitivity using the Matsuda Index.
Time Frame: 16 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are reported from the time the subjects sign the consent form until the completion of the study which includes baseline, medication ramp, exercise intervention, and follow up assessments. The total duration of the study for each subject is approximately 1 year.
Description: AEs are reported in real time by close research coordinator and participant interaction. They are graded according to intensity and causality and reported to the IRB in the appropriate amount of time. AEs were grouped according to body system such as musculoskeletal or gastrointestinal and reported together.
Arm/Group | Metformin | Placebo, Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/55
Other Adverse Events (participants affected / at risk) | 17/54 | 6/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=54) | Placebo, Sugar Pill (N=55)
Nausea, Diarrhea, Flatulence (Gastrointestinal disorders) | 17 (18) | 1 (1)
Musculoskeletal Pain or Injury (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT02308228/Prot_SAP_000.pdf
  • Informed Consent Form (2014-02-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT02308228/ICF_001.pdf